CLINICAL TRIAL: NCT00279279
Title: PREPARE - Primary Prevention Parameters Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 223
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Tachycardia, Ventricular; Implantable Cardioverter Defibrillator (ICD); Fibrillation, Ventricular; Syncope
Keywords: Implantable cardioverter defibrillator (ICD); Sudden Cardiac Death; Primary Prevention
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Syncope; Death, Sudden, Cardiac

INTERVENTIONS:
Device: Implanted Device

SUMMARY:
The purpose of this study is to test specific device programming in patients without a previous history of a life-threatening, abnormally fast heartbeat who are implanted with a Medtronic ICD (Implantable Cardioconverter Defibrillator) or ICD with CRT (Cardiac Resynchronozation Therapy) device. The information learned from this study could be used to guide physicians in future ICD or CRT device programming.

ELIGIBILITY:
Inclusion Criteria:

Patient is a candidate for a non-replacement Medtronic ICD device from the Marquis family or has had a non-replacement Medtronic Marquis based ICD system implanted within the previous 6 months and has not had any appropriately treated spontaneous VT/VF episodes during that time.

Exclusion Criteria:

Patient has history of spontaneous sustained symptomatic ventricular arrhythmias.

If patient has had an electrophysiology test in the past, and has sustained inducible VT <180 bpm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2003-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Demonstrate that patients programmed using a prescribed set of parameters have a lower rate of cardiac syncope, symptoms of fast heart rate, VT/VF events and cardioversion or defibrillation shocks compared to patients programmed per physician discretion

SECONDARY OUTCOMES:
Evaluate the percentage of inappropriate VT/VF detections
characterize the true incidence of VT/VF detections
therapy efficacy
time to first inappropriate VT/VF detection
incidence of untreated but monitored VT
programming changes
deaths and cardiovascular adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wilkoff, M.D, Principal Investigator — The Cleveland Clinic
Locations (32):
- United States (31):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - San Diego, California
  - San Pablo, California
  - Newark, Delaware
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Merrit Island, Florida
  - Columbus, Georgia
  - Maywood, Illinois
  - Rockford, Illinois
  - Topeka, Kansas
  - Portland, Maine
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Paterson, New Jersey
  - Buffalo, New York
  - New York, New York
  - Columbus, Ohio
  - Elyria, Ohio
  - Bethlehem, Pennsylvania
  - Lancaster, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Amarillo, Texas
  - Kirkland, Washington
  - Morgantown, West Virginia
- San Juan, Puerto Rico

REFERENCES:
- [Derived] van Gelder IC, Phan HM, Wilkoff BL, Brown ML, Rogers T, Peterson BJ, Birgersdotter-Green UM. Prognostic significance of atrial arrhythmias in a primary prevention ICD population. Pacing Clin Electrophysiol. 2011 Sep;34(9):1070-9. doi: 10.1111/j.1540-8159.2011.03124.x. Epub 2011 May 23. PMID 21605131
- [Derived] Wilkoff BL, Williamson BD, Stern RS, Moore SL, Lu F, Lee SW, Birgersdotter-Green UM, Wathen MS, Van Gelder IC, Heubner BM, Brown ML, Holloman KK; PREPARE Study Investigators. Strategic programming of detection and therapy parameters in implantable cardioverter-defibrillators reduces shocks in primary prevention patients: results from the PREPARE (Primary Prevention Parameters Evaluation) study. J Am Coll Cardiol. 2008 Aug 12;52(7):541-50. doi: 10.1016/j.jacc.2008.05.011. PMID 18687248